CLINICAL TRIAL: NCT01923935
Title: A Phase 2, Open-label, Prospective, Multicenter Study to Evaluate the Efficacy of Intravenous Busulfan and Melphalan as a Conditioning Regimen in Patients With Multiple Myeloma Undergoing Autologous Stem Cell Transplantation
Brief Title: Busulfan and Melphalan Conditioning in Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Je-Jung Lee, Professor, Chonnam National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KFDA20120110139
Record Dates: First submitted 2013-08-09; First posted 2013-08-16 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma, busulfan, melphalan,transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — Busulfan; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BUSULFEX®, Alkeran® (Experimental): BUSULFEX® 3.2 mg/kg/day iv once daily over 3 hours (day-6~day-4)
  Alkeran® 70 mg/m2/day iv once daily over 30 minutes (day-3~day-2)
  Interventions: Drug: BUSULFEX®; Drug: Alkeran®

INTERVENTIONS:
Drug: BUSULFEX® — BUSULFEX® 3.2 mg/kg/day iv once daily over 3 hours (day-6~day-4)
Drug: Alkeran® — Alkeran® 70 mg/m2/day iv once daily over 30 minutes (day-3~day-2)

SUMMARY:
The purpose of this study is to determine whether intravenous busulfan and melphalan as a conditioning regimen is effective in the treatment of multiple myeloma undergoing autologous stem cell transplantation.

DETAILED DESCRIPTION:
Title

* A phase 2, open-label, prospective, multicenter study to evaluate the efficacy of intravenous busulfan and melphalan as a conditioning regimen in patients with multiple myeloma (MM) undergoing autologous stem cell transplantation (ASCT)

Principal Investigator

* Je-Jung Lee (Chonnam National University Hwasun Hospital)

Co-investigators

* Hyeon Seok Eom (National Cancer Center)
* Kihyun Kim (Samsung Medical Center)
* Chang Ki Min (Seoul St. Mary's Hospital)
* Soo Jung Kim (Severance Hospital)
* Sung Soo Yoon (Seoul National University Hospital)
* Jae Hoon Lee (Gachon University Gil Hospital)
* Yeung-Chul Mun (Ewha Womans University Mokdong Hospital)

Duration

* 2 years

Study phase

* Phase II

Patients

* Patients with multiple myeloma who undergo autologous stem cell transplantation

Objectives(end points)

* Primary objective:

  1. Treatment response up to 2 months after ASCT
  2. Safety and toxicity (frequency of grade 3 or worse toxicities) of the conditioning regimen
* Secondary objective:

  1. Progression free survival (PFS)
  2. Overall survival (OS)

Total patients

* Initial 105 evaluable patients
* Complete Response (CR) rate of 200mg/m2 melphalan conditioning chemotherapy followed by ASCT in patients with newly diagnosed MM was about 26% and CR rate of busulfan and melphalan conditioning chemotherapy followed by ASCT in patients with newly diagnosed MM was about 40%. If the CR rate of busulfan and melphalan conditioning chemotherapy followed by ASCT is more than 40%, this combination will be accepted as active conditioning regimen that may be worth for investigating in phase III trial. But, if the CR rate of this regimen is lower than 26%, this has not a merit than 200mg/m2 melphalan conditioning chemotherapy. Based upon the above assumption, this trial was designed by using Simon's optimal two-stage testing procedure. Assuming a target level of interest, p1=0.4, and a lower activity level, p0=0.26 and drop rate 0.1. Initially 44 patients will be accrued. If 13 or more CR rate were observed, the trial will be continued. Accrual will be planned to a total of 105 patients, If total 35 or more patients were assessed as CR, busulfan and melphalan conditioning regimen will be accepted as active regimen, This design provides probability ≤ 0.05 of accepting drugs worse than p0 and probability ≤ 0.20 of rejecting drugs better than p1.if we assume that drop-out rate is 10%, total accrual patient will be 105

Treatment Schedule

* Busulfan 3.2 mg/kg/day iv once daily over 3 hours(day-6 ~ day-4)
* Melphalan 70 mg/m2/day iv once daily over 30 minutes(day-3 ~ day-1). If Creatinine Clearance (mL/min) < 50, reduce to 50 mg/m2. If Creatinine Clearance (mL/min) < 30, excluded from the this trial

Informed consent

* Written informed consent must be obtained before any study-specific screening procedures are performed

Screening

* Baseline assessments should be made within 28 days before treatment start:

  1. Demographic data (date of birth and sex)
  2. Eastern Cooperative Oncology Group performance status
  3. Vital signs and physical examination (including height, and weight)
  4. Medical history (including previous diseases/treatments and concomitant diseases/ treatments)
  5. Hematology - complete blood counts with differential count examination
  6. Serum electrolytes (Na, K, Cl, Ca, phosphorus)
  7. Serum lactate dehydrogenase
  8. Hepatitis B virus/hepatitis C virus/HIV serology (If serologic tests were conducted within 6 months prior to screening, retests are not required)
  9. Serum Beta2-microglobulin
  10. Quantitative serum M-protein (Serum protein electrophoresis), including immunofixation or immune electrophoresis
  11. Quantitative urine M-protein in 24 hrs urine (Urine protein electrophoresis), including immunofixation or immune electrophoresis
  12. Serum free light chain assay
  13. Creatinine clearance if increased serum creatinine
  14. ECG
  15. multigated radionuclide angiography or 2D ECHO
  16. Chest X-ray, Radiographic skeletal survey including skull, pelvis, vertebral column and long bones
  17. Bone marrow aspiration and biopsy with chromosome study, and flow cytometry or immunohistochemistry

Assessment

* Primary outcome measure

  1. To evaluate the objective responses after ASCT, the guidelines from the International Myeloma Working (IMW) Group uniform response criteria will be used
  2. Response Criteria for Multiple Myeloma the guidelines from the IMW Group uniform response criteria + Add for criteria of near CR (Immunofixation positive CR)
  3. Serum free light chain study will be added at the every evaluation of response
  4. To confirm the stringent complete response (sCR) after ASCT, flow cytometry or immunohistochemistry will be used
  5. NCI Common Toxicity Criteria for Adverse Effects version 4.0 will be used for the examination of toxicities
* Secondary outcome measure

  1. PFS will be defined from the time of ASCT to the time of first sign of disease progression or death
  2. OS will be defined as the period from the time of ASCT to the date of the last follow-up or death from any cause

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of MM
* Symptomatic MM
* Age 20 - 65 years
* The MM patients who performed the stem cell collection with appropriate stem cell counts, cluster of differentiation 34 positive cells more than 2 x 10^6 /kg
* Eastern Cooperative Oncology Group 0 - 2
* The MM patients who received induction chemotherapy regardless of types of induction
* Patient has measurable disease when the patients started the primary induction therapy, defined as follows: Measurable disease is defined as serum M-protein more than 1 g/dL, urine M-protein more than 200 mg/24 hours, or free light chain more than 100 mg/L
* Adequate liver functions before ASCT Transaminase less than 3 x upper normal value Bilirubin less than 2 x upper normal value
* Adequate hematological function - Platelet count more than 50,000 /microliter, hemoglobin more than 8 g / dL but, Prior red blood cell transfusion or recombinant human erythropoietin use is allowed, absolute neutrophil count more than 1,000 / microliter
* Expected survival: 6 months or more
* Informed consent

Exclusion Criteria:

* Systemic amyloid light chain amyloidosis, smoldering multiple myeloma or monoclonal gammopathy of undetermined significance
* Patient with plasma cell leukemia
* Patients who received an extensive radiation therapy within 4 weeks
* Patient is known to be Human Immunodeficiency Virus positive
* Patient has known clinically active Hepatitis B or C
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions Uncontrolled or severe cardiovascular disease, including myocardial infarction, within 6 months of enrollment, New York Heart Association Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis History of significant neurological or psychiatric disorders including dementia or seizures Active uncontrolled infection Active ulcers detected at gastroscopy Other serious medical illnesses
* Known hypersensitivity to any of the study drugs or its ingredients concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Treatment response up to 2 months after ASCT | 2 months later after last patent received ASCT
  1. To evaluate the objective responses after ASCT, the guidelines from the International Myeloma Working (IMW) Group uniform response criteria will be used.
  2. Serum free light chain study will be added at the every evaluation of response.
  3. To confirm the stringent complete response (sCR) after ASCT, flow cytometry or immunohistochemistry will be used
  Response Criteria for Multiple Myeloma:
  the guidelines from the IMW Group uniform response criteria + Add for criteria of near CR (Immunofixation positive CR)
Safety and toxicity (frequency of grade 3 or worse toxicities) of the conditioning regimen | 2 months later after last patent received ASCT
  NCI Common Toxicity Criteria for Adverse Effects version 4.0 will be used for the examination of toxicities.

SECONDARY OUTCOMES:
Progression free survival(PFS) | 2 months later after last patient received ASCT
  PFS will be defined from the time of ASCT to the time of first sign of disease progression or death.
Overall survival (OS) | 2 months later after last patient received ASCT
  OS will be defined as the period from the time of ASCT to the date of the last follow-up or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Je-Jung Lee, M.D., Ph.D., Principal Investigator — Chonnam National University Hospital
Locations (8):
- South Korea (8):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Gachon University Gil Hospital, Namdong-gu, Incheon
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Samsung Medical Center, Gangnam-gu, Seoul
  - Seoul National University Hospital, Jongno-gu, Seoul
  - Ewha Womans University Mokdong Hospital, Mokdong, Seoul
  - Seoul St. Mary's hospital, Seocho-gu, Seoul
  - Severance Hospital, Seodaemun-gu, Seoul

REFERENCES:
- [Background] McElwain TJ, Powles RL. High-dose intravenous melphalan for plasma-cell leukaemia and myeloma. Lancet. 1983 Oct 8;2(8354):822-4. doi: 10.1016/s0140-6736(83)90739-0. PMID 6137651
- [Background] Selby PJ, McElwain TJ, Nandi AC, Perren TJ, Powles RL, Tillyer CR, Osborne RJ, Slevin ML, Malpas JS. Multiple myeloma treated with high dose intravenous melphalan. Br J Haematol. 1987 May;66(1):55-62. doi: 10.1111/j.1365-2141.1987.tb06890.x. PMID 3593657
- [Background] Barlogie B, Tricot G, Anaissie E, Shaughnessy J, Rasmussen E, van Rhee F, Fassas A, Zangari M, Hollmig K, Pineda-Roman M, Lee C, Talamo G, Thertulien R, Kiwan E, Krishna S, Fox M, Crowley J. Thalidomide and hematopoietic-cell transplantation for multiple myeloma. N Engl J Med. 2006 Mar 9;354(10):1021-30. doi: 10.1056/NEJMoa053583. PMID 16525139
- [Background] Attal M, Harousseau JL, Stoppa AM, Sotto JJ, Fuzibet JG, Rossi JF, Casassus P, Maisonneuve H, Facon T, Ifrah N, Payen C, Bataille R. A prospective, randomized trial of autologous bone marrow transplantation and chemotherapy in multiple myeloma. Intergroupe Francais du Myelome. N Engl J Med. 1996 Jul 11;335(2):91-7. doi: 10.1056/NEJM199607113350204. PMID 8649495
- [Background] Fermand JP, Ravaud P, Chevret S, Divine M, Leblond V, Belanger C, Macro M, Pertuiset E, Dreyfus F, Mariette X, Boccacio C, Brouet JC. High-dose therapy and autologous peripheral blood stem cell transplantation in multiple myeloma: up-front or rescue treatment? Results of a multicenter sequential randomized clinical trial. Blood. 1998 Nov 1;92(9):3131-6. PMID 9787148
- [Background] Child JA, Morgan GJ, Davies FE, Owen RG, Bell SE, Hawkins K, Brown J, Drayson MT, Selby PJ; Medical Research Council Adult Leukaemia Working Party. High-dose chemotherapy with hematopoietic stem-cell rescue for multiple myeloma. N Engl J Med. 2003 May 8;348(19):1875-83. doi: 10.1056/NEJMoa022340. PMID 12736280
- [Background] Blade J, Rosinol L, Sureda A, Ribera JM, Diaz-Mediavilla J, Garcia-Larana J, Mateos MV, Palomera L, Fernandez-Calvo J, Marti JM, Giraldo P, Carbonell F, Callis M, Trujillo J, Gardella S, Moro MJ, Barez A, Soler A, Font L, Fontanillas M, San Miguel J; Programa para el Estudio de la Terapeutica en Hemopatia Maligna (PETHEMA). High-dose therapy intensification compared with continued standard chemotherapy in multiple myeloma patients responding to the initial chemotherapy: long-term results from a prospective randomized trial from the Spanish cooperative group PETHEMA. Blood. 2005 Dec 1;106(12):3755-9. doi: 10.1182/blood-2005-03-1301. Epub 2005 Aug 16. PMID 16105975
- [Background] Fermand JP, Katsahian S, Divine M, Leblond V, Dreyfus F, Macro M, Arnulf B, Royer B, Mariette X, Pertuiset E, Belanger C, Janvier M, Chevret S, Brouet JC, Ravaud P; Group Myelome-Autogreffe. High-dose therapy and autologous blood stem-cell transplantation compared with conventional treatment in myeloma patients aged 55 to 65 years: long-term results of a randomized control trial from the Group Myelome-Autogreffe. J Clin Oncol. 2005 Dec 20;23(36):9227-33. doi: 10.1200/JCO.2005.03.0551. Epub 2005 Nov 7. PMID 16275936
- [Background] Barlogie B, Kyle RA, Anderson KC, Greipp PR, Lazarus HM, Hurd DD, McCoy J, Moore DF Jr, Dakhil SR, Lanier KS, Chapman RA, Cromer JN, Salmon SE, Durie B, Crowley JC. Standard chemotherapy compared with high-dose chemoradiotherapy for multiple myeloma: final results of phase III US Intergroup Trial S9321. J Clin Oncol. 2006 Feb 20;24(6):929-36. doi: 10.1200/JCO.2005.04.5807. Epub 2006 Jan 23. PMID 16432076
- [Background] Alexanian R, Barlogie B, Tucker S. VAD-based regimens as primary treatment for multiple myeloma. Am J Hematol. 1990 Feb;33(2):86-9. doi: 10.1002/ajh.2830330203. PMID 2301376
- [Background] Barlogie B, Jagannath S, Desikan KR, Mattox S, Vesole D, Siegel D, Tricot G, Munshi N, Fassas A, Singhal S, Mehta J, Anaissie E, Dhodapkar D, Naucke S, Cromer J, Sawyer J, Epstein J, Spoon D, Ayers D, Cheson B, Crowley J. Total therapy with tandem transplants for newly diagnosed multiple myeloma. Blood. 1999 Jan 1;93(1):55-65. PMID 9864146
- [Background] Samson D, Gaminara E, Newland A, Van de Pette J, Kearney J, McCarthy D, Joyner M, Aston L, Mitchell T, Hamon M, et al. Infusion of vincristine and doxorubicin with oral dexamethasone as first-line therapy for multiple myeloma. Lancet. 1989 Oct 14;2(8668):882-5. doi: 10.1016/s0140-6736(89)91549-3. PMID 2571813
- [Background] Sirohi B, Powles R, Mehta J, Raje N, Kulkarni S, Ramiah V, Saso R, Horton C, Bhagwati N, Singhal S, Treleaven J. Complete remission rate and outcome after intensive treatment of 177 patients under 75 years of age with IgG myeloma defining a circumscribed disease entity with a new staging system. Br J Haematol. 1999 Dec;107(3):656-66. doi: 10.1046/j.1365-2141.1999.01744.x. PMID 10583272
- [Background] Goldschmidt H, Hegenbart U, Wallmeier M, Hohaus S, Haas R. Factors influencing collection of peripheral blood progenitor cells following high-dose cyclophosphamide and granulocyte colony-stimulating factor in patients with multiple myeloma. Br J Haematol. 1997 Sep;98(3):736-44. doi: 10.1046/j.1365-2141.1997.2783095.x. PMID 9332333
- [Background] Barlogie B, Alexanian R, Dicke KA, Zagars G, Spitzer G, Jagannath S, Horwitz L. High-dose chemoradiotherapy and autologous bone marrow transplantation for resistant multiple myeloma. Blood. 1987 Sep;70(3):869-72. PMID 3304465
- [Background] Jagannath S, Vesole DH, Glenn L, Crowley J, Barlogie B. Low-risk intensive therapy for multiple myeloma with combined autologous bone marrow and blood stem cell support. Blood. 1992 Oct 1;80(7):1666-72. PMID 1391937
- [Background] Moreau P, Facon T, Attal M, Hulin C, Michallet M, Maloisel F, Sotto JJ, Guilhot F, Marit G, Doyen C, Jaubert J, Fuzibet JG, Francois S, Benboubker L, Monconduit M, Voillat L, Macro M, Berthou C, Dorvaux V, Pignon B, Rio B, Matthes T, Casassus P, Caillot D, Najman N, Grosbois B, Bataille R, Harousseau JL; Intergroupe Francophone du Myelome. Comparison of 200 mg/m(2) melphalan and 8 Gy total body irradiation plus 140 mg/m(2) melphalan as conditioning regimens for peripheral blood stem cell transplantation in patients with newly diagnosed multiple myeloma: final analysis of the Intergroupe Francophone du Myelome 9502 randomized trial. Blood. 2002 Feb 1;99(3):731-5. doi: 10.1182/blood.v99.3.731. PMID 11806971
- [Background] Garban F, Attal M, Michallet M, Hulin C, Bourhis JH, Yakoub-Agha I, Lamy T, Marit G, Maloisel F, Berthou C, Dib M, Caillot D, Deprijck B, Ketterer N, Harousseau JL, Sotto JJ, Moreau P. Prospective comparison of autologous stem cell transplantation followed by dose-reduced allograft (IFM99-03 trial) with tandem autologous stem cell transplantation (IFM99-04 trial) in high-risk de novo multiple myeloma. Blood. 2006 May 1;107(9):3474-80. doi: 10.1182/blood-2005-09-3869. Epub 2006 Jan 5. PMID 16397129
- [Background] Moreau P, Milpied N, Mahe B, Juge-Morineau N, Rapp MJ, Bataille R, Harousseau JL. Melphalan 220 mg/m2 followed by peripheral blood stem cell transplantation in 27 patients with advanced multiple myeloma. Bone Marrow Transplant. 1999 May;23(10):1003-6. doi: 10.1038/sj.bmt.1701763. PMID 10373065
- [Background] Mansi J, da Costa F, Viner C, Judson I, Gore M, Cunningham D. High-dose busulfan in patients with myeloma. J Clin Oncol. 1992 Oct;10(10):1569-73. doi: 10.1200/JCO.1992.10.10.1569. PMID 1403036
- [Background] Bensinger WI, Rowley SD, Demirer T, Lilleby K, Schiffman K, Clift RA, Appelbaum FR, Fefer A, Barnett T, Storb R, Chauncey T, Maziarz RT, Klarnet J, McSweeney P, Holmberg L, Maloney DG, Weaver CH, Buckner CD. High-dose therapy followed by autologous hematopoietic stem-cell infusion for patients with multiple myeloma. J Clin Oncol. 1996 May;14(5):1447-56. doi: 10.1200/JCO.1996.14.5.1447. PMID 8622058
- [Background] Alegre A, Lamana M, Arranz R, Fernandez-Villalta MJ, Tomas JF, Figuera A, Camara R, Steegman JL, Casado F, Requena MJ, et al. Busulfan and melphalan as conditioning regimen for autologous peripheral blood stem cell transplantation in multiple myeloma. Br J Haematol. 1995 Oct;91(2):380-6. doi: 10.1111/j.1365-2141.1995.tb05307.x. PMID 8547079
- [Background] Fermand JP, Chevret S, Ravaud P, Divine M, Leblond V, Dreyfus F, Mariette X, Brouet JC. High-dose chemoradiotherapy and autologous blood stem cell transplantation in multiple myeloma: results of a phase II trial involving 63 patients. Blood. 1993 Oct 1;82(7):2005-9. PMID 8104534
- [Background] Ventura GJ, Barlogie B, Hester JP, Yau JC, LeMaistre CF, Wallerstein RO, Spinolo JA, Dicke KA, Horwitz LH, Alexanian R. High dose cyclophosphamide, BCNU and VP-16 with autologous blood stem cell support for refractory multiple myeloma. Bone Marrow Transplant. 1990 Apr;5(4):265-8. PMID 1970939
- [Background] Roussel M, Moreau P, Huynh A, Mary JY, Danho C, Caillot D, Hulin C, Fruchart C, Marit G, Pegourie B, Lenain P, Araujo C, Kolb B, Randriamalala E, Royer B, Stoppa AM, Dib M, Dorvaux V, Garderet L, Mathiot C, Avet-Loiseau H, Harousseau JL, Attal M; Intergroupe Francophone du Myelome (IFM). Bortezomib and high-dose melphalan as conditioning regimen before autologous stem cell transplantation in patients with de novo multiple myeloma: a phase 2 study of the Intergroupe Francophone du Myelome (IFM). Blood. 2010 Jan 7;115(1):32-7. doi: 10.1182/blood-2009-06-229658. Epub 2009 Nov 2. PMID 19884643
- [Background] Lahuerta JJ, Grande C, Blade J, Martinez-Lopez J, de la Serna J, Alegre A, Garcia LJ, Caballero D, de la Rubia J, Marin J, Perez-Lopez C, Sureda A, Escudero A, Cabrera R, Conde E, Garcia-Ruiz JC, Perez-Equiza K, Hernandez F, Palomera L, Leon A, Giraldo P, Solano C, Bargay J, San MJ; Spanish Multiple Myeloma Group. Myeloablative treatments for multiple myeloma: update of a comparative study of different regimens used in patients from the Spanish registry for transplantation in multiple myeloma. Leuk Lymphoma. 2002 Jan;43(1):67-74. doi: 10.1080/10428190210194. PMID 11908738
- [Background] Lahuerta JJ, Martinez-Lopez J, Grande C, Blade J, de la Serna J, Alegre A, Garcia-Larana J, Caballero D, Sureda A, de la Rubia J, Alvarez AM, Marin J, Escudero A, Conde E, Perez-Equiza K, Garcia Ruiz JC, Moraleda JM, Leon A, Bargay J, Cabrera R, Hernandez-Garcia MT, Diaz-Mediavilla J, Miguel JS. Conditioning regimens in autologous stem cell transplantation for multiple myeloma: a comparative study of efficacy and toxicity from the Spanish Registry for Transplantation in Multiple Myeloma. Br J Haematol. 2000 Apr;109(1):138-47. doi: 10.1046/j.1365-2141.2000.01979.x. PMID 10848793
- [Background] Carreras E, Rosinol L, Terol MJ, Alegre A, de Arriba F, Garcia-Larana J, Bello JL, Garcia R, Leon A, Martinez R, Penarrubia MJ, Poderos C, Ribas P, Ribera JM, San Miguel J, Blade J, Lahuerta JJ; Spanish Myeloma Group/PETHEMA. Veno-occlusive disease of the liver after high-dose cytoreductive therapy with busulfan and melphalan for autologous blood stem cell transplantation in multiple myeloma patients. Biol Blood Marrow Transplant. 2007 Dec;13(12):1448-54. doi: 10.1016/j.bbmt.2007.08.002. PMID 18022574
- [Background] Lahuerta JJ, Mateos MV, Martinez-Lopez J, Grande C, de la Rubia J, Rosinol L, Sureda A, Garcia-Larana J, Diaz-Mediavilla J, Hernandez-Garcia MT, Carrera D, Besalduch J, de Arriba F, Oriol A, Escoda L, Garcia-Frade J, Rivas-Gonzalez C, Alegre A, Blade J, San Miguel JF; Grupo Espanol de MM and Programa para el Estudio de la Terapeutica en Hemopatia Maligna Cooperative Study Groups. Busulfan 12 mg/kg plus melphalan 140 mg/m2 versus melphalan 200 mg/m2 as conditioning regimens for autologous transplantation in newly diagnosed multiple myeloma patients included in the PETHEMA/GEM2000 study. Haematologica. 2010 Nov;95(11):1913-20. doi: 10.3324/haematol.2010.028027. Epub 2010 Jul 27. PMID 20663944
- [Background] McDonald GB, Hinds MS, Fisher LD, Schoch HG, Wolford JL, Banaji M, Hardin BJ, Shulman HM, Clift RA. Veno-occlusive disease of the liver and multiorgan failure after bone marrow transplantation: a cohort study of 355 patients. Ann Intern Med. 1993 Feb 15;118(4):255-67. doi: 10.7326/0003-4819-118-4-199302150-00003. PMID 8420443
- [Background] Jones RJ, Lee KS, Beschorner WE, Vogel VG, Grochow LB, Braine HG, Vogelsang GB, Sensenbrenner LL, Santos GW, Saral R. Venoocclusive disease of the liver following bone marrow transplantation. Transplantation. 1987 Dec;44(6):778-83. doi: 10.1097/00007890-198712000-00011. PMID 3321587
- [Derived] Jung SH, Lee JJ, Kim JS, Min CK, Kim K, Choi Y, Eom HS, Joo YD, Kim SH, Kwak JY, Kang HJ, Lee JH, Lee HS, Mun YC, Moon JH, Sohn SK, Park SK, Park Y, Shin HJ, Yoon SS; Korean Multiple Myeloma Working Party. Phase 2 Study of an Intravenous Busulfan and Melphalan Conditioning Regimen for Autologous Stem Cell Transplantation in Patients with Multiple Myeloma (KMM150). Biol Blood Marrow Transplant. 2018 May;24(5):923-929. doi: 10.1016/j.bbmt.2018.01.004. Epub 2018 Jan 12. PMID 29339269